CLINICAL TRIAL: NCT00815334
Title: Efficacy of Endoscopic Subureteral Injection for Vesicoureteral Reflux in Adults With Decreased Bladder Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-094
Record Dates: First submitted 2008-12-28; First posted 2008-12-30 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-02

CONDITIONS: Vesicoureteral Reflux
Keywords: vesicoureteral reflux; low compliant bladder
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with decreased bladder compliance (Experimental): Patients who have decreased bladder compliance
  Interventions: Procedure: Endoscopic subureteric injection
- Patients with normal bladder compliance (Active Comparator): Patients who have normal bladder compliance
  Interventions: Procedure: Endoscopic subureteric injection

INTERVENTIONS:
Procedure: Endoscopic subureteric injection — Endoscopic subureteric injection for the treatment of vesicoureteral reflux using variable materials (polydimethylsiloxane, collagen, and dextranomer/hyaluronic acid copolymer)

SUMMARY:
Endoscopic subureteral injection for vesicoureteral reflux has become an established alternative to ureter reimplantation in children. Some recent studies suggest that ESI can be also a primary treatment option for VUR in adults. However, the experience with ESI in adults who have VUR associated with decreased bladder compliance is limited. We evaluated the efficacy of endoscopic subureteral injection treatment for vesicoureteral reflux in adults with decreased bladder compliance.

ELIGIBILITY:
Inclusion Criteria:

* Who is aged 18 and greater
* Who underwent endoscopic subureteral injection for vesicoureteral reflux

Exclusion Criteria:

* Medical records of whom is not evaluabe

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cure rate | 3, 12 months

SECONDARY OUTCOMES:
adverse events | 3, 12 months
predictive factor for cure | 3, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D., M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Choo MS, Hong B, Ji YH, Chung H, Choe JH, Park WH, Park T, Lee KS. Endoscopic treatment of vesicoureteral reflux with polydimethylsiloxane in adult women. Eur Urol. 2004 Jun;45(6):787-9. doi: 10.1016/j.eururo.2003.11.025. PMID 15149753
- [Background] Okeke Z, Fromer D, Katz MH, Reiley EA, Hensle TW. Endoscopic management of vesicoureteral reflux in women presenting with pyelonephritis. J Urol. 2006 Nov;176(5):2219-21. doi: 10.1016/j.juro.2006.07.076. PMID 17070296
- [Background] Puri P. Endoscopic correction of vesicoureteral reflux. Curr Opin Urol. 2000 Nov;10(6):593-7. doi: 10.1097/00042307-200011000-00010. PMID 11148731